CLINICAL TRIAL: NCT05610410
Title: Relationship Between Regulation of Peripheral and Intracoronary Microvascular Blood Flow in Patients With Ischemia and no Obstructive Coronary Arteries
Brief Title: Peripheral Microvascular Blood Flow in ANOCA
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Yolande Appelman, MD, PhD, FESC, VU University of Amsterdam
Other Study IDs: VUmc_2021.0615
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-06

CONDITIONS: ANOCA - Angina With Non-obstructive Coronary Arteries; HFpEF - Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with angina and no obstructive coronary arteries
  Interventions: Other: Laser speckle contrast analysis
- Patients with HFpEF
  Interventions: Other: Laser speckle contrast analysis

INTERVENTIONS:
Other: Laser speckle contrast analysis — Peripheral endothelial function assessment using Laser speckle contrast analysis and Peripheral reactive hyperemia assessment using EndoPAT
  Other Names: EndoPAT

SUMMARY:
An observational cross-sectional cohort study investigating whether peripheral endothelial function assessed using Laser speckle contrast analysis and coronary endothelial function measured with invasive coronary function testing are correlated in patients with angina and no obstructive coronary arteries.

DETAILED DESCRIPTION:
Rationale: Coronary endothelial dysfunction (CED) has been proposed to cause signs and symptoms of myocardial ischaemia in patients with angina but no obstructive coronary artery disease (INOCA) and has been proposed to play an important role in the pathophysiology of heart failure with preserved ejection fraction, as an element of the pro-inflammatory state causing cardiac functional and structural abnormalities in this syndrome. Research has shown that patients with coronary microvascular dysfunction (CMD) often present with echocardiographic signs of diastolic dysfunction combined with higher rates of detectable cardiac troponin and are at increased risk of developing HFpEF, indicating a major overlap in the complex pathophysiology underlying these syndromes. CED is associated with an increased risk of adverse cardiac events and currently can only be detected with invasive coronary function testing (ICFT).

However, it has been suggested that CED is a component of systemic endothelial dysfunction and is associated with endothelial dysfunction in other microvascular beds. The cutaneous microcirculation is suitable for microvascular function studies and has been shown to correlate with muscle microvascular function. The recently developed Laser speckle contrast analysis (LASCA) technique enables non-invasive monitoring of microvascular blood flow in superficial microvascular beds. In combination with iontophoresis of acetylcholine, nitroprusside and insulin, LASCA allows evaluation of peripheral microvascular endothelial and smooth muscle function. While LASCA is an established technique, the association between CED diagnosed with ICFT and an abnormal peripheral endothelial function measured by LASCA is currently unknown.

Objective: The primary objective of the study is to test whether peripheral endothelial function assessed using Laser speckle contrast analysis and CED measured with ICFT are correlated.

Study design: Observational cross-sectional cohort study.

Study population: 51 patients over the age of 18 with signs and symptoms of ischemia with no obstructive coronary arteries (INOCA) and a clinical indication for ICFT because of persistent angina without obstructive coronary artery disease and 58 patients with heart failure with preserved ejection fraction (HFpEF) and a clinical indication for ICFT.

Primary study endpoint: The main study end point is the difference in peripheral endothelial function between patients with and without CED measured with ICFT in the INOCA group and the HFpEF group.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Study participants do not benefit from participation in this study. The burden of this study is low. The aim is that study procedures will be performed within 24 hours of the elective ICFT and study participants do not have to come to the hospital for an additional visit. The total risks associated with participation are classified as being low, because the risks for adverse events and serious adverse events from a local and transient stimulus in skin are minimal. Iontophoresis of acetylcholine, nitroprusside and insulin does not cause any skin damage and the used dosages are very small and as such, the stimuli do not cause any systemic effects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for elective invasive coronary function test (ICFT)
* Suited for one of the study groups:

  * Persistent angina, defined as symptoms of angina; or
  * HFpEF, diagnosed according to the European Society of Cardiology 2021 heart failure guidelines
* Absence of obstructive CAD, documented before inclusion, defined as

  * Coronary Computed Tomography Angiography (CCTA) - indicative of absence of obstructed coronary arteries, or
  * Coronary angiography (CAG) - <50% diameter stenosis (DS) in the epicardial coronary arteries or (fractional flow reserve (FFR) >0.80 or instant wave free ratio (iFR) >0.89)

Exclusion Criteria:

* Under 18 years of age
* Unable or unwilling to undergo ICFT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed to evaluate INOCA patients with a clinical indication of ICFT because of persistent angina without obstructive coronary artery disease and HFpEF patients with a clinical indication of ICFT.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Laser speckle contrast analysis (LASCA) | 35 minutes
  Peripheral microvascular function measured with Laser speckle contrast analysis (LASCA) between patients with non-obstructive coronary artery disease with and without Coronary endothelial dysfunction. LASCA measures microvasclar function non invasively by measure perfusion units (APU/mmHg.)

SECONDARY OUTCOMES:
EndoPAT | 15 minutes
  The relationship between microvascular reactivity measured using EndoPAT in patients with angina and non-obstructive coronary ateries (ANOCA) or heart failure with preserved ejection fraction (HFpEF). The EndoPAT displays the pulse amplitude response to ischemia, and automatically calculates the Reactive Hyperemia Index (RHI). RHI index measures post-ischemic vasodilatation, which is partly mediated by endothelium-derived nitric oxide (NO). RHI is calculated as the post-to-pre occlusion PAT-signal ratio in the index finger of the occlude arm, divided by the corresponding ratio from the contralateral, control arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, lcoation VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No